CLINICAL TRIAL: NCT01446068
Title: Comparison of Postprandial Inflammation in Lean and Obese Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Agroscope Liebefeld-Posieux Research Station ALP (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NUTRICHIP-1
Record Dates: First submitted 2011-09-29; First posted 2011-10-04 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Nutritional Intervention; Nutritional and Metabolic Diseases; Obesity
MeSH Terms: conditions — Nutritional and Metabolic Diseases; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lean Subjects (Experimental)
  Interventions: Dietary Supplement: High-fat meal
- Obese subjects (Experimental)
  Interventions: Dietary Supplement: High-fat meal

INTERVENTIONS:
Dietary Supplement: High-fat meal — Three caloric doses of high-fat meal (500, 1000, 1500 kcal)

SUMMARY:
The purpose of this study is to quantify the systemic inflammatory and metabolic response of lean subjects and obese subjects to the ingestion of three caloric doses of a high-fat meal.

ELIGIBILITY:
Inclusion Criteria for lean subjects:

* age 25-50
* 20<BMI<25
* waist circumference <94cm

Inclusion Criteria for obese subjects

* age-matched to healthy subjects
* 30<BMI<40
* waist circumference >102cm

Exclusion Criteria for lean and obese subjects:

* Physiological or psychological diseases
* Allergies to food or intolerance to high-fat meal
* Vegetarians
* Chronic intake of drugs
* Smokers
* Diabetes mellitus Type I and II
* Debilitating kidney diseases
* Debilitating liver diseases
* Clinically established coronary heart diseases
* Ingestion of vitamins or dietary supplements during the course of the study

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Interleukin-6 (serum) | 4h vs 0h
  A statistically-significant increase in serum Interleukin-6 is expected at 4h compared to 0h

SECONDARY OUTCOMES:
Glucose (serum) | 0h, 1h, 2h, 4h, 6h
Triglyceride (serum) | 0h, 1h, 2h, 4h, 6h
Insulin (serum) | 0h, 1h, 2h, 4h, 6h
high sensitivity C-Reactive Protein | 0h, 1h, 2h, 4h, 6h
HDL-cholesterol | 0h, 1h, 2h, 4h, 6h
Total cholesterol | 0h, 1h, 2h, 4h, 6h
Total cholesterol / HDL cholesterol | 0h, 1h, 2h, 4h, 6h
Interleukin-6 (serum) | 0h, 1h, 2h, 4h, 6h
Glucagon-like-protein-1 (serum) | 0h, 1h 2h, 4h, 6h
Endotoxin (serum) | 0h, 1h, 2h, 4h, 6h

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Laederach, MD, Study Director — Inselspital University of Berne; Katrin Bolanz, PhD, Principal Investigator — Agroscope Liebefeld-Posieux ALP Research Station; Flurina Schwander, M.Sc., Principal Investigator — Agroscope Liebefeld-Posieux ALP Research Station; Caroline Buri, MD, Principal Investigator — Inselspital University of Berne
Locations (2):
- Switzerland (2):
  - Agroscope Liebefeld-Posieux ALP Research Station, Bern, Canton of Bern
  - University Hospital Inselspital, Berne, Bern, Canton of Bern

REFERENCES:
- [Derived] Schwander F, Kopf-Bolanz KA, Buri C, Portmann R, Egger L, Chollet M, McTernan PG, Piya MK, Gijs MA, Vionnet N, Pralong F, Laederach K, Vergeres G. A dose-response strategy reveals differences between normal-weight and obese men in their metabolic and inflammatory responses to a high-fat meal. J Nutr. 2014 Oct;144(10):1517-23. doi: 10.3945/jn.114.193565. Epub 2014 May 8. PMID 24812072